CLINICAL TRIAL: NCT04037670
Title: Assessment of the Efficacy of SASI Bypass in Super Obese Patients With BMI> 50 Kg/m2
Brief Title: Efficacy of SASI Bypass in Super Obese Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Sameh Emile, Lecturer of surgery, Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: mansoura101
Record Dates: First submitted 2019-07-28; First posted 2019-07-30 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SASI bypass (Experimental): Patients with super obesity underwent SASI bypass
  Interventions: Procedure: SASI bypass

INTERVENTIONS:
Procedure: SASI bypass — Sleeve gastrectomy with single loop anastomosis between gastric antrum and ileum, 3 meters away from ileocecal junction

SUMMARY:
Although previous studies investigated weight loss and improvement in comorbidities after SASI bypass, patients included in these studies had a BMI less than 50 Kg/m2. Therefore, the aim of the present study was to investigate the outcome of SASI bypass in patients with super obesity to assess the success of this novel bariatric procedure in this challenging group of patients in regards weight loss and improvement in associated comorbid conditions at 12 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients included to the present study were adult patients of both genders aging between 18 and 65 years with primary morbid obesity with BMI ≥50 kg/m2 with or without obesity-associated comorbidities such as hypertension, diabetes mellitus (DM), dyslipidemias, and gastroesophageal reflux disease (GERD).

Exclusion Criteria:

* Pregnant women.
* Patients unfit for general anasthesia (ASA 4, 5)
* Endocrine or psychiatric disorders.
* History of previous upper abdmominal laparotomy.
* Alcoholic addiction
* Liver cirrhosis
* Coagulopathy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-07-20 (Actual); Study Completion 2019-07-20 (Actual)

PRIMARY OUTCOMES:
percentage of excess weight loss | at 12 months of follow-up
  [preoperative weight - weight at 12 months]/preoperative excess weight X 100

SECONDARY OUTCOMES:
Resolution of diabetes mellitus | at 12 months of follow-up
  number of patients with fasting plasma glucose level <110 mg/dL or HbA1C level <6% without hypoglycemic medication

CONTACTS AND LOCATIONS:
Overall Officials: Sameh H Emile, M.D., Principal Investigator — Mansoura University
Locations (1):
- Mansoura university hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided